CLINICAL TRIAL: NCT01939899
Title: An Open-label, Multicenter, Phase 2 Study of Oral IXAZOMIB (MLN9708) in Adult Patients With Relapsed and/or Refractory Follicular Lymphoma
Brief Title: Phase 2 Study of Oral IXAZOMIB in Adult Participants With Relapsed and/or Refractory Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16017; 2013-002302-32 (EudraCT Number); U1111-1164-7551 (Other: WHO); 166547 (Registry Identifier: HC-CTD); REec-2016-2137 (Registry Identifier: REec); 13/EM/0373 (Registry Identifier: NRES)
Record Dates: First submitted 2013-08-28; First posted 2013-09-11 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Follicular Lymphoma
Keywords: MLN9708; Lymphoma; IXAZOMIB
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IXAZOMIB (Experimental): Ixazomib 4, 5.3 and 7 milligram (mg), orally, once on Days 1, 8 and 15 in a 28 day treatment cycle followed by a rest period of 13 days, for up to Cycle 29 or until disease progression or unacceptable toxicity at lead-in phase for participants with NHL. After completion of lead-in phase, participants will continue into Phase 2. Participants in Phase 2 will receive Ixazomib at RP2D dose, orally, once weekly on Days 1, 8 and 15 in a 28 day treatment cycle followed by a rest period of 13 days , for up to Cycle 29 or until disease progression or unacceptable toxicity in Phase 2 for participants with RRFL.
  Interventions: Drug: IXAZOMIB

INTERVENTIONS:
Drug: IXAZOMIB — Each 28-day treatment cycle will include oral administration of IXAZOMIB on Days 1, 8, and 15 followed by a rest period of 13 days.
  Other Names: MLN9708

SUMMARY:
The primary purpose of this study is to evaluate the anti-tumor activity of oral Ixazomib as measured by overall response rate (ORR) in adult participants with relapsed and/or refractory follicular lymphoma (FL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years or older.
* Participants must have a pathologically confirmed diagnosis of non-Hodgkin lymphoma (NHL) (for the lead-in dose-finding phase) and FL (for phase 2).
* Participants must have radiographically or clinically measurable disease.
* Participants must be relapsed and/or refractory after at least 1 prior therapy (excluding radiation) with documented progressive disease at the time of enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to practice true abstinence.
* Male participants who agree to practice effective barrier contraception or agree to practice true abstinence.
* Voluntary written consent.
* Suitable venous access.
* Appropriate clinical laboratory values as defined in the protocol.
* Recovered from toxicities of prior anticancer therapy.
* If the trial proceeds to the second step on the basis of the tandem 2-step design, participants must be confirmed PSMB1 positive at the central laboratory before treatment.

Exclusion Criteria

* Peripheral neuropathy that is greater or equal to Grade 2 or Grade 1 with pain.
* Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period.
* Autologous stem cell transplant within 6 months before Day 1 of Cycle 1, or prior allogeneic stem cell transplant at any time.
* Major surgery within 14 days before the first dose of study drug.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
* Comorbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the participants inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Evidence of current uncontrolled cardiovascular conditions including uncontrolled hypertension, severe uncontrolled ventricular arrhythmias, unstable angina, New York Heart Association (NYHA) Class III or IV cardiac disease, or myocardial infarction within the past 6 months.
* Diarrhea greater than (>) Grade 1 on the basis of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) categorization.
* Systemic antineoplastic (including glucocorticoids > the equivalent of 15 mg of prednisone daily), experimental, or radiation therapy within 21 days before the first dose of study drug.
* Prior treatment with rituximab or other unconjugated antibody treatment within 42 days (21 days if clear evidence of progressive disease or immediate treatment is mandated).
* Treatment with radioimmunoconjugates or toxin immunoconjugates within 12 weeks before the first dosing of study treatment.
* Systemic treatment with strong inhibitors of Cytochrome P450 1A2 (CYP1A2) or Cytochrome P450 3A (CYP3A), or strong CYP3A inducers within 14 days before the first dose of IXAZOMIB - Ongoing systemic therapy with corticosteroids.
* Central nervous system (CNS) involvement that is clinically uncontrolled or newly diagnosed in the last 4 months.
* Ongoing or active systemic viral infection, known human immunodeficiency virus (HIV) positive, known active hepatitis B virus or known active hepatitis C virus.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease with the exception of nonmelanoma skin cancer or any completely resected carcinoma in situ.
* Platelet transfusions within 3 days before the 1st dose of study drug.
* Inability to swallow capsules, or inability or unwillingness to avoid taking anything by mouth except for water and prescribed medication for 2 hours before and 1 hour after dose of IXAZOMIB - Known allergy to boron or excipients in the formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (14):
- United States (4):
  - Boston, Massachusetts
  - New York, New York
  - Nashville, Tennessee
  - Houston, Texas
- Belgium (3):
  - Ghent
  - Leuven
  - Wilrijk
- Montreal, Quebec, Canada
- United Kingdom (6):
  - London
  - Manchester
  - Newcastle upon Tyne
  - Plymouth
  - Southampton
  - Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in the United States, Belgium, Canada, United Kingdom and Italy from 31 October 2013 to 23 March 2017.
Pre-assignment Details: Participants with follicular lymphoma (FL) prior to treatment were enrolled in this 2 phase study: Lead in dose finding phase in which maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of ixazomib was evaluated and Phase 2 proteasome subunit beta type-1 (PSMB1) was done to evaluate the safety, efficacy, tolerability of ixazomib.
Groups:
- Lead-in Dose Finding Phase: Ixazomib 4 mg: Ixazomib 4 milligram (mg), solution, orally, once on Day 1, 8, and 15 followed by 13 days of rest in a 28-days treatment cycle for a maximum of 29 cycles, or progressive disease (PD) or the start of alternate therapies during lead-in dose finding in non-hodgkin lymphoma (NHL) participants.
- Lead-in Dose Finding Phase: Ixazomib 5.3 mg: Ixazomib 5.3 mg, solution, orally, once on Day 1, 8, and 15 followed by 13 days of rest in a 28-days treatment cycle for a maximum of 29 cycles, or PD or the start of alternate therapies during lead-in dose finding in NHL participants.
- Lead-in Dose Finding Phase: Ixazomib 7.0 mg: Ixazomib 7 mg, solution, orally, once on Day 1, 8, and 15 followed by 13 days of rest in a 28-days treatment cycle for a maximum of 29 cycles, or PD or the start of alternate therapies during lead-in dose finding in NHL participants.
- Phase 2: PSMB1 Positive: Ixazomib RP2D mg, solution, orally, once weekly on Day 1, 8, and 15 followed by 13 days of rest in a 28-days treatment cycle for a maximum of 29 cycles, or PD or the start of alternate therapies during phase 2 finding in relapsed Or refractory follicular lymphoma (RRFL) participants.
- Phase 2: PSMB1 Negative: Ixazomib RP2D mg, solution, orally, once weekly on Day 1, 8, and 15 followed by 13 days of rest in a 28-days treatment cycle for a maximum of 29 cycles, or PD or the start of alternate therapies during phase 2 finding in RRFL participants.
Period: Lead-in Dose Finding Phase
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Started | 3 | 7 | 6 | 0 | 0
Completed | 1 | 0 | 1 | 0 | 0
Not Completed | 2 | 7 | 5 | 0 | 0
Not completed — Death | 0 | 3 | 1 | 0 | 0
Not completed — Disease Progression | 2 | 4 | 3 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Period: Phase 2
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Started | 0 | 0 | 0 | 12 | 1
Completed | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 11 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 9 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who had received at least 1 dose of ixazomib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative | Total
Number analyzed (Participants) | 3 | 7 | 6 | 12 | 1 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (6.56) | 57.9 (11.13) | 64.3 (7.71) | 64.7 (11.73) | 79.0 (NA) — Standard deviation could not be calculated since only 1 participant was analyzed. | 64.2 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The safety population included all enrolled participants who had received at least 1 dose of ixazomib.
  Participants
    Female | 1 | 1 | 1 | 4 | 1 | 8
    Male | 2 | 6 | 5 | 8 | 0 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The safety population included all enrolled participants who had received at least 1 dose of ixazomib.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 3 | 7 | 6 | 12 | 0 | 28
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Population: The safety population included all enrolled participants who had received at least 1 dose of ixazomib.
  participants
    Belgium | 1 | 2 | 3 | 3 | 0 | 9
    Canada | 0 | 1 | 2 | 0 | 0 | 3
    United Kingdom | 0 | 3 | 1 | 2 | 0 | 6
    Italy | 0 | 0 | 0 | 5 | 0 | 5
    United States | 2 | 1 | 0 | 2 | 1 | 6
Smoking classification [Count of Participants; unit: Participants] — Population: The safety population included all enrolled participants who have received at least 1 dose of ixazomib.
  Participants
    Never smoked | 2 | 4 | 5 | 7 | 1 | 19
    Current smoker | 0 | 2 | 0 | 0 | 0 | 2
    Ex-smoker | 1 | 1 | 1 | 5 | 0 | 8
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The safety population included all enrolled participants who have received at least 1 dose of ixazomib.
  centimeter (cm) | 170.0 (7.04) | 175.0 (11.50) | 169.2 (9.11) | 168.8 (6.70) | 157.5 (NA) — Standard deviation could not be calculated since only 1 participant was analyzed. | 170.1 (8.77)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The safety population included all enrolled participants who have received at least 1 dose of ixazomib.
  kilogram (kg) | 76.1 (11.27) | 85.8 (20.72) | 85.3 (10.95) | 78.7 (13.54) | 82.4 (NA) — Standard deviation could not be calculated since only 1 participant was analyzed. | 81.6 (14.45)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the investigator using the international Working Group criteria for participants CR: disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Baseline up to Day 15 Cycle 29 (approximately up to Day 802) or until PD or the start of alternate therapies
Population: The response-evaluable population included all participants who received at least 1 dose of ixazomib, had measurable disease at baseline, and had at least 1 post baseline disease assessment.
Measure: Number; unit: participants
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Number analyzed (Participants) | 3 | 5 | 5 | 12 | 1
participants
  CR | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 1 | 0
  Stable Disease (SD) | 1 | 2 | 2 | 4 | 0
  PD | 2 | 3 | 3 | 7 | 1

2. Secondary Outcome: Lead-in Dose Finding Phase: Recommended Phase 2 Dose (RP2D)
Time Frame: Baseline up to Cycle 1 Day 28
Population: The dose limiting toxicity (DLT)- evaluable population included all participants who received all Cycle 1 doses of ixazomib and had completed Cycle 1 safety procedures, or experience a DLT in Cycle 1 in the lead-in dose finding phase of the study.
Measure: Number; unit: mg
Groups:
- Lead-in Dose Finding Phase: All Participants: Ixazomib 5.3 mg, solution, orally, once on Day 1, 8, and 15 followed by 13 days of rest in a 28-days treatment cycle for a maximum of 29 cycles, or PD or the start of alternate therapies during lead-in dose finding in NHL participants.
Arm/Group | Lead-in Dose Finding Phase: All Participants
Number analyzed (Participants) | 16
mg | 5.3

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first dose of study treatment to the date of first documented PD or death. Participants without documentation of PD will be censored at the date of last response assessment that is SD or better. Participants without response assessment will be censored at the date of first dose.
Time Frame: Time from the date of first dose of study treatment to the date of first documented PD or death (approximately up to Day 802)
Population: The modified intent-to-treat (mITT) population included all participants who received at least 1 dose of ixazomib in the phase 2 portion of the study or who received at least 1 dose of ixazomib and are treated at the RP2D in the lead-in dose finding phase of the study.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Lead-in Dose Finding: Ixazomib 5.3 mg (RP2D): Ixazomib 5.3 mg, solution, orally, once on Day 1, 8, and 15 followed by 13 days of rest in a 28-days treatment cycle for a maximum of 29 cycles, or PD or the start of alternate therapies during lead-in dose finding in NHL participants.
Arm/Group | Lead-in Dose Finding: Ixazomib 5.3 mg (RP2D) | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Number analyzed (Participants) | 7 | 12 | 1
months | 1.9 [1.68 to 3.71] | 2.4 [1.87 to 11.50] | NA [NA to NA] — Median and confidence interval could not be calculated since only 1 participant was analyzed.

4. Secondary Outcome: Phase 2: Rate of Disease Control
Description: Rate of disease control is defined as percentage of participants who achieved a SD or better for greater than or equal to (>=) 6 months.
Time Frame: Baseline or until occurrence of disease progression, unacceptable toxicities, or discontinuation of study due to any other reasons (approximately up to Day 805)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Number analyzed (Participants) | 12 | 1
percentage of participants | 16.7 [2.09 to 48.41] | NA [NA to NA] — Confidence interval could not be calculated since no participant had rate of disease control.

5. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from the date of first dose of study treatment to the date of the first documentation of a PR or better response in a participant who responded.
Time Frame: Time from the date of first dose of study treatment to the date of first documented PR or better response or death (approximately up to Day 802)
Population: The response-evaluable population included all participants who received at least 1 dose of ixazomib, had measurable disease at baseline, and had at least 1 post baseline disease assessment. Participants who were evaluable for this given measure at a given time point were included for this assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
days |  |  |  | 560 |

6. Secondary Outcome: Duration of Response (DOR)
Description: The DOR is defined as the time from the date of first documentation of a response to the date of first documented PD. Responders without documentation of PD will be censored at the date of last response assessment. DOR was categorized as CR+PR and CR.
Time Frame: Time from the date of first documentation of a response to the date of first documented PD (approximately up to Day 802)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
months |  |  |  | 0.0328542094 |

7. Secondary Outcome: Phase 2: Number of Participants With Response Rates in PSMB1 Positive and PSMB1 Negative
Time Frame: Baseline up to occurrence of disease progression, unacceptable toxicities, or discontinuation of study due to any other reasons (approximately up to Day 802)
Population: The biomarker population included all participants positive or negative for the PSMB1 biomarker and where the assay has passed quality control. Data will be derived from a baseline blood sample.
Measure: Number; unit: participants
Arm/Group | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Number analyzed (Participants) | 12 | 1
participants | 12 | 1

8. Secondary Outcome: Number of Participants Experiencing 1 or More Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to 30 days after last dose of study drug (approximately up to Day 832)
Population: The safety population included all enrolled participants who had received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
Number analyzed (Participants) | 3 | 7 | 6 | 12 | 1
participants
  TEAE | 3 | 7 | 6 | 11 | 1
  SAE | 1 | 3 | 4 | 4 | 1

9. Secondary Outcome: Lead-in Dose Finding Phase: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Cycle 1, Days 1 and 15 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The plasma pharmacokinetic (PK) analysis population included all participants enrolled in the lead-in dose finding phase that had sufficient dosing data and ixazomib concentration-time data. The PK analysis population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg
Number analyzed (Participants) | 3 | 7 | 6
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 141.3333 (52.27173) | 103.4717 (57.53181) | 121.1167 (69.07212)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 3
  Cycle 1 Day 15 | 124.2667 (71.01840) | 144.0667 (105.15884) | 152.0667 (102.71131)

10. Secondary Outcome: Lead-in Dose Finding Phase: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Time Frame: Cycle 1, Days 1 and 15 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The PK analysis population included all participants enrolled in the lead-in dose finding phase that had sufficient dosing data and ixazomib concentration-time data. The PK analysis population where data at specified time points was available.
Measure: Median (Full Range); unit: hour
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg
Number analyzed (Participants) | 3 | 7 | 6
hour
  Cycle 1 Day 1 | 1.0000 [0.500 to 1.500] | 1.0000 [0.500 to 1.500] | 1.0500 [1.000 to 3.750]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 3
  Cycle 1 Day 15 | 1.0000 [0.500 to 2.000] | 0.7500 [0.467 to 1.520] | 1.0000 [0.500 to 1.500]

11. Secondary Outcome: Lead-in Dose Finding Phase: AUC(0-168): Area Under the Plasma Concentration-time Curve From Time 0 to 168 Hours Postdose for Ixazomib
Time Frame: Cycle 1, Days 1 and 15 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The PK analysis set where Cycle 1 Day 1 and 15 assessment were available. The PK analysis population included all participants enrolled in the lead-in dose finding phase that had sufficient dosing data and ixazomib concentration-time data. The PK analysis population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg
Number analyzed (Participants) | 3 | 7 | 6
hour*nanogram per milliliter (h*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 7 | 6
  Cycle 1 Day 1 | 1265.0000 (332.34019) | 1030.1429 (367.90326) | 1680.3333 (656.01240)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 3
  Cycle 1 Day 15 | 2440.0000 (272.21315) | 2007.0000 (986.30117) | 3120.0000 (2503.83706)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to Cycle 29)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Lead-in Dose Finding Phase: Ixazomib 4 mg | Lead-in Dose Finding Phase: Ixazomib 5.3 mg | Lead-in Dose Finding Phase: Ixazomib 7.0 mg | Phase 2: PSMB1 Positive | Phase 2: PSMB1 Negative
All-Cause Mortality (participants affected / at risk) | 0/3 | 3/7 | 1/6 | 0/12 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/7 | 4/6 | 4/12 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6 | 11/12 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in Dose Finding Phase: Ixazomib 4 mg (N=3) | Lead-in Dose Finding Phase: Ixazomib 5.3 mg (N=7) | Lead-in Dose Finding Phase: Ixazomib 7.0 mg (N=6) | Phase 2: PSMB1 Positive (N=12) | Phase 2: PSMB1 Negative (N=1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in Dose Finding Phase: Ixazomib 4 mg (N=3) | Lead-in Dose Finding Phase: Ixazomib 5.3 mg (N=7) | Lead-in Dose Finding Phase: Ixazomib 7.0 mg (N=6) | Phase 2: PSMB1 Positive (N=12) | Phase 2: PSMB1 Negative (N=1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 6 (10) | 5 (17) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (5) | 3 (4) | 3 (7) | 5 (11) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 4 (10) | 5 (16) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (5) | 3 (3) | 2 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (6) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (11) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (4) | 3 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.